CLINICAL TRIAL: NCT03206996
Title: Treatment for Auditory Hyper-Reactivity Behavior in Children With Autism Using Exposure and Response Prevention Principles
Brief Title: Exposure Therapy for Auditory Sensitivity in Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201601664
Record Dates: First submitted 2017-06-26; First posted 2017-07-02 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Sensory Disorders; Autism; Autism Spectrum Disorder; Autism With High Cognitive Abilities; Autistic Behavior; Hyperacusis
Keywords: autism; sensory over-responsiveness; auditory hyper-sensitivity; auditory processing; exposure therapy; exposure and response prevention; cognitive behavior therapy; occupational therapy
MeSH Terms: conditions — Sensation Disorders; Autistic Disorder; Autism Spectrum Disorder; Child Development Disorders, Pervasive; Hyperacusis | interventions — Implosive Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Single-subjects design (baseline, treatment and follow-up)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Child Interventional (Experimental): A 12 week patient-centered modified E/RP protocol for up to 5 participants with ASD and auditory hyper-reactivity. E/RP protocols will include face-to-face treatment sessions as well as the provision of home programs. Treatment fidelity checklists will be utilized each session to ensure that each participant receive the same general protocol/treatment process
  Interventions: Behavioral: Exposure therapy; Behavioral: Psycho-education; Behavioral: Caregiver education/home program development
- Parental Interventional (Experimental): A 12 week patient-centered modified E/RP protocol for up to 5 participants with ASD and auditory hyper-reactivity. E/RP protocols will include face-to-face treatment sessions as well as the provision of home programs. Treatment fidelity checklists will be utilized each session to ensure that each participant receive the same general protocol/treatment process
  Interventions: Behavioral: Caregiver education/home program development

INTERVENTIONS:
Behavioral: Exposure therapy — The therapist, child and family collaborate to set short and long term goals, develop the exposure hierarchy and Subjective Units of Distress (SUD) scale and design their "challenge" activities (i.e., exposures). The exposure hierarchy lists activities in ascending order from minimal exposure/minimally difficult (e.g, toilet is not flushed and bathroom door is closed while child walks by) to maximum exposure/maximally difficult (e.g., toilet is flushed repeatedly while child is inside the stall with the door closed). Treatment begins with exposure to activities on the lower end of the hierarchy, with adjustments as indicated, to present stimuli that provide a "just-right" level of difficulty as indicated by the participant's SUD level and therapists clinical judgment. Participants communicate the level of difficulty using their individualized SUD scale. Additionally, the child and family complete home exercises with exposures.
  Other Names: cognitive behavioral therapy; exposure and response prevention; systematic desensitization
  Arms: Child Interventional
Behavioral: Psycho-education — Child and caregiver receive education and training will be provided to improve the participant's self-awareness of his/her behavioral and emotional response to auditory stimuli, his/her ability to self-report anxiety/emotional response levels, as well as his/her ability to identify useful arousal level modulation/coping strategies. During this phase, the child, caregiver and therapist will collaborate to identify the participant's Subjective Units of Distress Scale (SUD) from 0-10 with each level defined, particularly for what levels are tolerable or intolerable.
  Arms: Child Interventional
Behavioral: Caregiver education/home program development — Parents will be provided with education on home programs to facilitate treatment gains. Home programs will be designed specifically for each participant. Parent education and home programs are provided either concurrently or after the exposure phase for the family to apply these methods to other settings. Home programs can continue as a maintenance program after treatment has ended. At the end of the treatment phase, the study team will conduct the following assessments for a third time: (1) the Sensory Profile, a clinical tool commonly used in OT to assess parent reports of sensory processing difficulties in children, (2) Parent Stress Index - 4 to evaluate stress related to parent-child interactions, and (3) the Modified Khalfa Hyper-acusis Questionnaire to assess the level of hyper-sensitivity to sound.

SUMMARY:
Auditory hyper-reactivity affects up to 66% of children with autism spectrum disorder (ASD) and has been linked to greater stress and anxiety for children and their families. Exposure and Response Prevention (E/RP) is highly effective for reducing obsessive/compulsive behaviors in children with both OCD and ASD. This study is the first to assess the feasibility and efficacy of E/RP for auditory sensory hyper-reactivity in ASD.

DETAILED DESCRIPTION:
Sensory processing difficulties have been well documented in children with Autism Spectrum Disorder (ASD). In fact, "hyper- or hypo-reactivity to sensory input" has recently been added to the diagnostic criteria of this disorder. Hyper-reactivity features are particularly disruptive to children's abilities to engage in everyday activities and pose a significant problem for patients and their families. In children with high functioning pervasive developmental disorder, hyper-sensitivity is associated with symptoms of anxiety and depression. For sensory processing difficulties, children with ASD are primarily referred to Occupational Therapy (OT) services for treatment. These patients are also often seen by mental health professionals to address related disorders such as anxiety, ADHD and behavior problems. Currently, there are no evidence based approaches for specifically addressing auditory hyper-reactivity in ASD. Exposure and response prevention (E/RP), derived from systematic desensitization, is highly effective at reducing avoidance behaviors associated with phobias and obsessive and compulsive disorder (OCD). In mental healthcare settings, ER/P has been shown to be effective for reducing compulsive behaviors in children with OCD and concurrent ASD. E/RP has also been piloted for treating restricted, repetitive behaviors in ASD and demonstrates good feasibility. E/RP may also be useful for reducing aversive responses to auditory stimuli in children with ASD. Occupational Therapists (OT) are the primary service for providing treatment for sensory processing and arousal level modulation difficulties in children with ASD. Thus, OTs are potentially well suited to provide an E/RP aimed at reducing sensory hyper-reactivity in ASD. This study will investigate the feasibility and efficacy of utilizing an E/RP approach for treating auditory hyper-reactivity in ASD.

ELIGIBILITY:
Inclusion Criteria of children:

* autism spectrum disorders (ASD) diagnosis with symptoms of auditory hyper-sensitivity/reactivity.
* verbal communication skills for utilizing the Subjective Units of Distress (SUD) scale (no cut-off for IQ).

Exclusion Criteria of children

* behavioral diagnosis of Oppositional Defiant Disorder or Conduct Disorder
* history of child abuse that is related to sound sensitivity

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Participant Subjective Unit of Distress (SUD) Level | weekly for approximately 20 weeks from intake to exit
  The Subjective Unit of Distress (SUD) scale is a 0-10 scale used for the child and/or caregiver to report level of distress (i.e., pain, stress, anxiety, discomfort) before, during and/or after exposures to stimuli. We expect that SUDS levels will decrease over time indicating improved ability to tolerate auditory stimuli.

SECONDARY OUTCOMES:
Parent Stress Index | intake, end of baseline, end of treatment and exit (up to 4 times over approximately 20 weeks from intake to exit)
  As an exploratory secondary outcome measure we will look for changes in scores on the parent Stress Index, a 36 item (5 point Likert scale response) parent report that is useful for identifying potential issues regarding the child's or parent's behavior and level of stress. It is also useful for designing treatment plans, setting goals, follow-up and evaluating pre-/post- treatment outcomes.
Spence Child Anxiety Scale | intake, end of baseline, end of treatment and exit (up to 4 times over approximately 20 weeks from intake to exit)
  As an exploratory secondary outcome measure we will look for changes in scores on the Spence Children's Anxiety Scale (SCAS). The SCAS child-report is a 45 item questionnaire and the SCAS Parent-Report is a 39 item questionnaires with 4-point Likert scale responses. Both forms assess six domains of anxiety including generalized anxiety, panic/agoraphobia, social phobia, separation anxiety, obsessive compulsive disorder and physical injury fears.
Modified Khalfa Hyperacusis Questionnaire | intake, end of baseline, end of treatment and exit (up to 4 times over approximately 20 weeks from intake to exit)
  As an exploratory secondary outcome measure we will look for changes in scores on the Modified Khalfa Hyperacusis Questionnaire, a brief 20 item (3-point Likert scale) questionnaire to screen for auditory hypersensitivity (hyper-acusis).
Autism Symptoms | intake (week 1) and exit (final session approximately 20 weeks after intake)
  As an exploratory secondary outcome measure we will look for changes in scores on the Autism Diagnostic Observation Schedule - 2 (ADOS-2) and the Autism Spectrum Rating Scales (ASRS). The ADOS-2 is a play-based assessment that provides direct observation of the child's behavior and the ASRS is a norm-referenced, 71 item Likert scale parent questionnaire that identifies symptoms and behaviors across the autism spectrum.
Sensory Profile | intake, end of baseline, end of treatment and exit (up to 4 times over approximately 20 weeks from intake to exit)
  As an exploratory secondary outcome measure we will look for changes in scores on the Sensory Profile-2. The Sensory Profile is an 86 item (5-point Likert scale) parent questionnaire (age 3-14) or Adolescent/adult questionnaire (ages 15 and above) that is used to evaluate how sensory processing and behaviors in a child compare to peers; norm-referenced on the following sensory sections: auditory, visual, touch, movement, body position, oral; behavioral sections: conduct, social/emotional and attention; as well as the following quadrants: seeking, avoiding, sensitivity and registration.

CONTACTS AND LOCATIONS:
Overall Officials: Tana Carson, PhD, Principal Investigator — Adjunct Associate Research Professor
Locations (2):
- United States (2):
  - UF Health Child and Adolescent Psychiatry/Medical Psychology, Gainesville, Florida
  - University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: Undecided